CLINICAL TRIAL: NCT04441333
Title: Usability, Safety and Efficacy of AspivixTM, an Atraumatic Innovative Uterine Cervical Traction Device: a Pilot Phase Followed by a Comparative Study (Pilot)
Brief Title: Usability, Safety and Efficacy of AspivixTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspivix SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Aspivix_IUD2019_Pilot
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: IUD Insertion

STUDY DESIGN:
Intervention Model Description: Pilot study: single-arm non-comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AspivixTM cervical vacuum tenaculum (Experimental): Traction of the cervix for IUD insertion using the AspivixTM cervical vacuum tenaculum.
  Interventions: Device: AspivixTM cervical vacuum tenaculum

INTERVENTIONS:
Device: AspivixTM cervical vacuum tenaculum — Traction of the cervix for IUD insertion using the AspivixTM cervical vacuum tenaculum

SUMMARY:
Limited mobility of the uterine cervix and alignment with the vaginal canal is often required during insertion of an intrauterine contraceptive device (IUD). Currently, the available instruments are traumatic tenacula, which could cause pain and bleeding and therefore represent an obstacle for certain patients to pursue their medical follow-up.

AspivixTM is a new device, which enables atraumatic traction of the cervix while respecting its specific semi-circular anatomic shape through a system powered by a vacuum chamber.

The aim of our pilot study is to assess the usability, safety and efficacy of the device.

Note: Study is made of 2 phases (pilot phase followed by a comparative phase). Details regarding comparative study is registered separately.

ELIGIBILITY:
Inclusion Criteria:

* Participants older than 18 years
* Participants presenting at the outpatient clinic for Mirena IUD insertion.
* Participants able to provide informed consent as documented by signature with at least 24 hours of reflection time
* Good understanding of written and oral speaking used at the centre where the study will be carried out.

Exclusion Criteria:

* Participants who are contraindicated for the insertion of the IUD Mirena
* Participants under use of excessive alcohol, narcotics or benzodiazepines prior to procedure
* Participants who do not wish to be informed of a chance discovery
* Participant receiving anaesthetics prior to IUD insertion procedure
* Participants on anticoagulant medication
* Participants under use of an analgesic
* Previous cervical operation
* Severe vaginal bleeding
* Participant previously enrolled in this study
* Cervix diameter smaller than 26 mm
* Mullerian anomalies with two cervices
* Nabothian cyst
* Cervical myomas
* Cervical condylomas
* Squamous intraepithelial lesion (Cervical dysplasia)
* Cervical endometriosis
* Cervical tears
* A well exposed cervix and / or well aligned vaginal and cervical canals where no traction is required for IUD insertion
* Other cervical abnormalities (cervical polyp, cervical lesion, or irregularity) which may contraindicate or complicate IUD insertion
* Large ectopy, for which it is not possible to find a suitable location near the ectopy where native tissue is present
* Large scar tissue, for which it is not possible to find a suitable location near the scar where native tissue is present

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Usability and efficacy from the practitioner's perspective: questionnaire | Right after the use of the device (right after the end of the procedure to insert the IUD).
  The practitioner will assess the usability and efficacy of the Investigational Device using a 5 point Likert 'Usability and Efficacy Questionnaire'.

SECONDARY OUTCOMES:
Participant's reported pain: Visual Analogue Scale | Before the procedure, during speculum insertion, during AspivixTM vacuum application, during application of cervical traction, during IUD insertion, during AspivixTM release, 5 minutes after the end of the procedure
  Participant's reported pain will be assessed by the patient using a 100-point Visual Analogue Scale (VAS) at specific steps during IUD insertion Minimum and maximum values range from 0 to 100, the higher score being the better outcome.
Assessment of patient's satisfaction: questionnaire | Right after the use of the device (right after the end of the procedure to insert the IUD).
  5 point Likert 'Patient Satisfaction Questionnaire' Minimal to maximal values range from 1 to 5, 1 meaning "disagree" and 5 "agree".
The number of placement attempts before traction can be applied | During the procedure to insert the IUD which should last less than 5 minutes.
  The number of placement attempts before traction of the cervix can be applied will be recorded
The number of spontaneous releases during traction | During the procedure to insert the IUD which should last less than 5 minutes.
  The number of spontaneous releases during traction of the cervix will be recorded
Assessment of bleeding | During the procedure to insert the IUD which should last less than 5 minutes.
  To assess bleeding, every buffer will be weighted, and the blank weight subtracted. Weight in mg will be reported in the case report form.
Assessment of adverse events | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by documenting adverse events (description of the adverse events, number of participants)
Assessment of device deficiencies | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by documenting device deficiencies (description of the deficiency)
Identification of new risks | During the procedure to insert the IUD which should last less than 5 minutes.
  Safety of the procedure will be assessed by identifying and documenting any new risk.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Mathevet, Prof., Principal Investigator — DFME CHUV Lausanne
Locations (1):
- Department Women, Mother & Child, University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legardeur H, Masiello-Fonjallaz G, Jacot-Guillarmod M, Mathevet P. Safety and Efficacy of an Atraumatic Uterine Cervical Traction Device: A Pilot Study. Front Med (Lausanne). 2021 Dec 23;8:742182. doi: 10.3389/fmed.2021.742182. eCollection 2021. PMID 35004719